CLINICAL TRIAL: NCT02349958
Title: Clinical Trial of Intraperitoneal Hyperthermic Chemotherapy Using Cisplatin, Mitomycin, and Adriamycin in Peritoneal Surface Malignancies Also Known as Hyperthermic Intraperitoneal Chemotherapy.
Brief Title: Clinical Trial of Intraperitoneal Hyperthermic Chemotherapy
Acronym: HIPEC/IPHC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bay Area Gynecology Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIPEC
Record Dates: First submitted 2014-12-22; First posted 2015-01-29 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer; Uterine Cancer; Mesotheliomas; Gastrointestinal Cancers; Cervical Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Uterine Neoplasms; Mesothelioma; Gastrointestinal Neoplasms; Uterine Cervical Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ovarian peritoneal (Other): CDDP Cisplatin 75 mg/m2 @T0 Ovarian peritoneal fallopian tube Uterine
  Interventions: Device: HIPEC: CDDP 75 mg/m2 @T0
- Appendix Psuedomyxoma (Other): MMC Mitomycin 30mg @ T0, 10mg @ T45min 50 mg/m2 @T0 Appendix Psuedomyxoma colorectal small bowel
  Interventions: Device: HIPEC: MMC 30mg @ T0, 10mg @ T45min
- Gastric and Pancreato-biliary (Other): MMC Mitomycin + CDDP Cisplatin 30mg @ T0, 10mg @ T45min 50 mg/m2 @T0
  Interventions: Device: HIPEC: MMC + CDDP 30mg @ T0, 10mg @ T45min 50 mg/m2 @T0
- Mesothelioma and Sarcoma (Other): CDDP Cisplatin + Doxorubicin 50 mg/m2 @T0 15 mg/m2 @T0
  Interventions: Device: HIPEC: CDDP+ Doxorubicin 50 mg/m2 @T0 15 mg/m2 @T0

INTERVENTIONS:
Device: HIPEC: MMC 30mg @ T0, 10mg @ T45min — MMC 30mg @ T0, 10mg @ T45min for Appendix, Psuedomyxoma, colorectal, small bowel
  Other Names: HIPEC
  Arms: Appendix Psuedomyxoma
Device: HIPEC: MMC + CDDP 30mg @ T0, 10mg @ T45min 50 mg/m2 @T0 — Gastric and Pancreato-biliary HIPEC: MMC + CDDP 30mg @ T0, 10mg @ T45min
  Arms: Gastric and Pancreato-biliary
Device: HIPEC: CDDP 75 mg/m2 @T0 — Ovarian/peritoneal/fallopian tube, Uterine CDDP 75 mg/m2 @T0
  Arms: Ovarian peritoneal
Device: HIPEC: CDDP+ Doxorubicin 50 mg/m2 @T0 15 mg/m2 @T0 — CDDP+ Doxorubicin 50 mg/m2 @T0 15 mg/m2 @T0 Mesothelioma and Sarcoma
  Arms: Mesothelioma and Sarcoma

SUMMARY:
To determine treatment response to surgical debulking and intra-operative Intraperitoneal Hyperthermic Chemotherapy (IPHC) in patients with the following malignancies:

Gynecologic cancers (ovarian, primary peritoneal or fallopian tube, and uterine/cervical cancers).

Mesotheliomas. GI cancers (Gallbladder, liver, small intestine, pancreas, stomach, colon, appendix).

To monitor the toxicities and complications of this treatment regimen. To measure treatment related QOL changes after IPHC.

DETAILED DESCRIPTION:
PSC is, by definition, a metastatic stage of malignancy. Ovarian cancer, and clinically identical entities (fallopian tube and primary peritoneal cancer) are most commonly found to spread as a PSC. These diseases seldom spread outside of the peritoneal cavity even after multiple recurrences. Therefore, clinical experience with IPHC is nearly all from ovarian (and related) cancers.

Ovarian cancer is the leading cause of death from a gynecologic malignancy in the United States. There are approximately 26,000 new cases and 14,500 deaths annually. Primary peritoneal and fallopian tube carcinomas are significantly less frequent than ovarian cancer, but outcomes and treatments are identical. The recommended initial treatment for these diseases is to perform a staging operation with aggressive debulking of tumor. These patients then receive intravenous, or intraperitoneal, taxane and platinum-based chemotherapy to treat the residual disease. This treatment yields overall median survivals of approximately 37 months in patients that were suboptimally debulked (residual tumor, >1.0 cm in diameter) and 49 months in those with optimally debulked disease (residual tumor, 1.0 cm in diameter). Overall, approximately 75% of those with Stage II-IV ovarian cancer will respond to their initial adjuvant chemotherapy and 50% are clinically without evidence of disease at the completion of their adjuvant chemotherapy cycles. However, 50% of these patients would have persistent disease identified at the time of a second look laparotomy. Of those with a negative second look laparotomy, 50% will experience a recurrence of their disease. Second Look Laparotomy is a controversial choice for patients who have no evidence of disease by non-invasive means after their primary treatment. It appears that some patients may benefit in Progression Free Survival (PFS) when complete cytoreduction of residual disease is possible, but no randomized trial exists to prove 5 year survival benefit. Patients that recur after their initial adjuvant chemotherapy will generally die from their disease, as salvage therapy has not been very effective. At the present time, the initial adjuvant regimen consists of a platinum and paclitaxel-based regimen as the standard therapy for these patients. Cisplatin was originally used for the intravenous regimens and continues to be used for intraperitoneal (IP) therapy. In fact, the GOG has now made IP cisplatin a part of the standard adjuvant regimen for optimally debulked ovarian cancer patients. This shift was based on the analysis of three randomized trials that support the IP cisplatin route. Patients in this Gynecologic Oncology Group (GOG) trial underwent optimal cytoreductive surgery and were randomly assigned to a control group receiving intravenous paclitaxel and intravenous cisplatin or to an experimental group receiving intravenous paclitaxel on day 1, intraperitoneal cisplatin on day 2, and intraperitoneal paclitaxel on day 8. At a median follow-up of 50 months, there was a statistically significant prolongation of median progression-free survival and overall survival in the intraperitoneal treatment group (a benefit of 5.5 and 15.9 months, respectively). This represented a 25 percent reduction in the risk of death. This 15.9-month improvement in median overall survival is one of the longest survival benefits ever observed for a new therapy in gynecologic oncology.

Uterine disease may be divided into cancer of the cervix, and cancer of the corpus, which behave quite differently, even when compared by similar histology subtype.

Corpus epithelial cancer is a common Gynecologic malignancy, with 41,200 projected 2006 cases resulting in an estimated 3,750 deaths. This is by far more prevalent than ovarian-related cancers, and usually quite curable at early stage. Approximately 10-15% of cases, however, are found outside of the uterus (Stage III or IV) at presentation. These cases have a poor outcome, with only 30% of Stage III patients (disease spread to regional lymph nodes, peritioneal fluid, or pelvis) and less than 5% of Stage IV (spread to abdominal cavity) surviving 5 years. Recurrent disease occurs in approximately 29% of Stage I patients Patients with recurrence ultimately die of disease, and often are treated medically with a survival of 13-15 months. However, recent retrospective studies have shown that patients with recurrent disease can reasonably be offered surgery, with better outcomes from complete cytoreduction. Median survival times are range from 35 to 43.0 months, for those with small or no residual tumor, compared to 10-13.5 months for those patients with gross residual disease. Sarcomas of the uterus are rare, representing only 2-5% of all corpus cancers. These are staged and treated much like high-grade epithelial cancer, but these patients have poorer survivals when compared to similar stage for common histologic subtypes. Early stage patients survive to five years less than 50% of the time. Those with more advanced disease has a 0-20% five-year survival (median survival 4-26 months). Studies on these diseases have been subjected to low numbers, due to the rarity of disease, and few conclusions can be drawn. However, surgical debulking is thought to be probably beneficial.

Cervical cancers are expected to account for 9,710 cases with 3,700 deaths in 2006. The disease is often discovered at early stage, confined to the cervix (Stage I) and is often curable. Cure rates in these patients are directly related to cervical disease volume, with survivals ranging from 71-90%. However, between 14.4-25.6% of patients with early disease will recur after initial radiation or surgical therapy, within 3 years. Recurrent disease is usually in the pelvis, and treatable fairly successfully with surgical exenteration. Extrapelvic spread of disease is only confined to the peritoneal cavity in 8% of cases, but treatment of these patients is currently considered futile.

OBJECTIVES

To determine Overall Survival for surgical debulking and intra-operative Intraperitoneal Hyperthermic Chemotherapy (IPHC) in patients with the following malignancies:

Gynecologic cancers (ovarian, primary peritoneal or fallopian tube, and uterine/cervical cancers). Mesotheliomas. GI cancers (Gallbladder, liver, small intestine, pancreas, stomach, colon, appendix).

To determine the number of Grade III and Grade IV CTCAE v4.03 toxicities and complications of this treatment regimen.

To measure treatment related QOL changes after IPHC.

ELIGIBILITY:
PATIENT ELIGIBILITY

Presumptive clinical diagnosis of a peritoneal surface cancer (PSC) prior to surgery, with no metastases outside of the abdomen.

Patients must have a performance status of 0, 1, or 2.

Patients must have adequate:

Bone marrow function: absolute neutrophil count more than or equal to 1500 and platelet count more than or equal to 100,000 Renal function: creatinine less than or equal to 1.5 mg/dl Hepatic function: bilirubin less than or equal 1.5times upper limit of normal, SGOT and alkaline phosphatase less than or equal 2.5 times upper limit of normal range Patients must have signed an informed consent. Patients of childbearing potential must have a negative serum pregnancy test prior to study entry and be practicing an effective form of contraception.

Patients are at least 18 years of age, and under 75 years of age.

At the time of surgery, operative assessment and frozen section diagnosis of one of the following:

Primary ovarian cancer (POC) with Stage IC or greater stage Recurrent or persistent ovarian cancer (ROC) Ovarian cancer patients who desire Consolidation Chemotherapy (CC). These patients would ordinarily choose to have 12 cycles of Taxol given after standard first-line surgery and chemotherapy, and instead choose one course of IPHC as their CC.

Uterine malignancy of the corpus, or cervix with primary tumor Stage IIIA or greater, or recurrent tumor confined to the abdomen.

Metastatic mesothelioma or sarcoma confined to the abdomen. Recurrent or primary gastrointestinal cancer, with regional spread confined to the peritoneal cavity

PATIENT INELIGIBILITY

Patients with known extra-abdominal disease, or unresected bulky abdominal retroperitoneal lymph nodes.

Patients with any evidence of another malignancy within the last five years (except non-melanoma skin cancer) Patients with a known sensitivity to cisplatin, Mitomycin C, or Adriamycin. Patients with significant co-morbid medical conditions that would prevent the patient from completing treatment on this protocol, per Investigator discretion.

Patients desiring future fertility.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-09; Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
measure treatment response to HIPEC and tumor debulking | 10 years
  To determine Overall Survival HIPEC and tumor debulking in patients with the following malignancies:
  Gynecologic cancers (ovarian, primary peritoneal or fallopian tube, and uterine/cervical cancers).
  GI cancers (Gallbladder, liver, small intestine, pancreas, stomach, colon, appendix).
  EVALUATION CRITERIA Postoperative monitoring of toxicity and treatment (Appendix I) CR, PR, stable disease and progressive disease will be monitored. The endpoints to be examined are increase or decrease in the size of measurable ascites, tumor, and tumor markers (CA-125, CA-19.9, or CEA).
  Performance status Quality of Life Physical examination

SECONDARY OUTCOMES:
Toxicity Monitoring | 10 Years
  1.2. To determine the number of Grade III and Grade IV CTCAE v4.03 toxicities and complications of this treatment regimen.

OTHER OUTCOMES:
QOL | 10 years
  1.3. To measure treatment related QOL changes after IPHC/ HIPEC

CONTACTS AND LOCATIONS:
Overall Officials: James Lilja, MD, Principal Investigator — Bay Area Gynecology Oncology
Locations (1):
- James Lilja, Los Gatos, California, United States